CLINICAL TRIAL: NCT02158533
Title: A Phase 3 Efficacy and Safety Study of ALKS 5461 for the Adjunctive Treatment of Major Depressive Disorder (the FORWARD-4 Study)
Brief Title: A Study of ALKS 5461 for the Treatment of Major Depressive Disorder (MDD) - the FORWARD-4 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK5461-205
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Alkermes; ALKS 5461; Samidorphan
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose (Experimental)
  Interventions: Drug: High Dose ALKS 5461
- Low Dose (Experimental)
  Interventions: Drug: Low Dose ALKS 5461
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: High Dose ALKS 5461 — Sublingual tablet, taken once daily (in addition to open-label treatment with a commercially available antidepressant)
  Other Names: ALKS 5461
  Arms: High Dose
Drug: Low Dose ALKS 5461 — Sublingual tablet, taken once daily (in addition to open-label treatment with a commercially available antidepressant)
  Other Names: ALKS 5461
  Arms: Low Dose
Drug: Placebo — Sublingual tablet, taken once daily (in addition to open-label treatment with a commercially available antidepressant)
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index (BMI) of 18.0 to 40.0 kg/m2, inclusive
* Agree to use an acceptable method of contraception for the duration of the study
* Have a Major Depressive Disorder (MDD) primary diagnosis
* Have no more than 2 inadequate responses to antidepressant therapy (ADT) in the current Major Depressive Episode (MDE)
* Additional criteria may apply

Exclusion Criteria:

* Have a current primary Axis-I disorder other than MDD
* Have used opioid agonists (eg, codeine, oxycodone, tramadol, morphine) or opioid antagonists (eg, naloxone, naltrexone) within 14 days
* Have received electroconvulsive therapy treatment within the last 2 years or received more than one course of electroconvulsive treatment during lifetime
* Have attempted suicide within the past 2 years
* Have a positive test for drugs of abuse
* Are pregnant, planning to become pregnant, or breastfeeding
* Have a history of intolerance, allergy, or hypersensitivity to buprenorphine or opioid antagonists (eg, naltrexone, naloxone)
* Have had a significant blood loss or blood donation within 60 days
* Additional criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (47):
- United States (40):
  - Alkermes Investigational Site, Birmingham, Alabama
  - Alkermes Investigational Site, Tucson, Arizona
  - Alkermes Investigational Site, Carson, California
  - Alkermes Investigational Site, National City, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Sherman Oaks, California
  - Alkermes Investigational Site, Torrance, California
  - Alkermes Investigational Site, Upland, California
  - Alkermes Investigational Site, Hartford, Connecticut
  - Alkermes Investigational Site, Norwich, Connecticut
  - Alkermes Investigational Site, Coral Springs, Florida
  - Alkermes Investigational Site, Gainesville, Florida
  - Alkermes Investigational Site, Lauderhill, Florida
  - Alkermes Investigational Site, Orlando, Florida
  - Alkermes, Investigational Site, Alpharetta, Georgia
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Joliet, Illinois
  - Alkermes Investigational Site, Skokie, Illinois
  - Alkermes Investigational Site, Newburgh, Indiana
  - Alkermes Investigational Site, Valparaiso, Indiana
  - Alkermes Investigational Site, Owensboro, Kentucky
  - Alkermes Investigational Site, Baltimore, Maryland
  - Alkermes Investigational Site, Berlin, New Jersey
  - Alkermes Investigational Site, Brooklyn, New York
  - Alkermes Investigational Site, Mount Kisco, New York
  - Alkermes Investigational Site, New York, New York
  - Alkermes Investigational Site, Staten Island, New York
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Allentown, Pennsylvania
  - Alkermes Investigational Site, Media, Pennsylvania
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Lincoln, Rhode Island
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, San Antonio, Texas
  - Alkermes Investigational Site, Woodstock, Vermont
  - Alkermes Investigational Site, Middleton, Wisconsin
- Australia (4):
  - Alkermes Investigational Site, Brisbane, Queensland
  - Alkermes Investigational Site, Towong, Queensland
  - Alkermes Investigational Site, Frankston, Victoria
  - Alkermes Investigational Site, Melbourne, Victoria
- Canada (3):
  - Alkermes Investigational Site, Penticton, British Columbia
  - Alkermes Investigational Site, Gatineau, Quebec
  - Alkermes Investigational Site, Québec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were diagnosed with major depressive disorder (MDD) and had an inadequate response to 1 or 2 adequate courses of treatment with a commercially available antidepressant therapy (ADT) during the current major depressive episode (MDE). All subjects continued ADT for the duration of the study.
Pre-assignment Details: This was a Sequential Parallel Comparison Design (SPCD) study comprised of 2 stages. In Stage 1 subjects were randomized to ALKS 5461 or placebo (2:2:9). In Stage 2 only placebo non-responders from Stage 1 were re-randomized to ALKS 5461 or placebo (1:1:1). One subject randomized to the PBO group in Stage 1 did not receive study drug.
Groups:
- Placebo S1: Randomized to placebo in Stage 1
- ALKS 5461 0.5mg/0.5mg S1: Randomized to ALKS 5461 0.5mg/0.5mg in Stage 1
- ALKS 5461 2mg/2mg S1: Randomized to ALKS 5461 2mg/2mg in Stage 1
- Placebo S2: Randomized to placebo in Stage 2
- ALKS 5461 0.5mg/0.5mg S2: Randomized to ALKS 5461 0.5mg/0.5mg in Stage 2
- ALKS 5461 2mg/2mg S2: Randomized to ALKS 5461 2mg/2mg in Stage 2
Period: Stage 1
Arm/Group | Placebo S1 | ALKS 5461 0.5mg/0.5mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 0.5mg/0.5mg S2 | ALKS 5461 2mg/2mg S2
Started | 265 | 59 | 60 | 0 | 0 | 0
Completed | 251 | 51 | 52 | 0 | 0 | 0
Not Completed | 14 | 8 | 8 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 4 | 7 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Failure to Meet Eligibility Criteria | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study visits | 1 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Placebo S1 | ALKS 5461 0.5mg/0.5mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 0.5mg/0.5mg S2 | ALKS 5461 2mg/2mg S2
Started (Subjects randomized in Stage 2 are a subset of those randomized to placebo in Stage 1.) | 0 | 0 | 0 | 56 | 56 | 56
Completed | 0 | 0 | 0 | 53 | 52 | 50
Not Completed | 0 | 0 | 0 | 3 | 4 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Psychiatrist decision to try new tx | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Non-adherence with study visits | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects randomized to Stage 1 (i.e., all subjects randomized during the study) who received ≥ 1 dose of study drug.
Groups:
- ALKS 5461 0.5mg/0.5mg S1: Randomized to ALKS 0.5mg/0.5mg in Stage 1
- ALKS 5461 2mg/2mg S1: Randomized to ALKS 5461 2/2 in Stage 1
- Total: Total of all reporting groups
Arm/Group | Placebo S1 | ALKS 5461 0.5mg/0.5mg S1 | ALKS 5461 2mg/2mg S1 | Total
Number analyzed (Participants) | 265 | 59 | 60 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (11.50) | 45.0 (13.89) | 46.2 (12.14) | 45.7 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 38 | 40 | 260
  Male | 83 | 21 | 20 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 7 | 4 | 44
  Not Hispanic or Latino | 232 | 52 | 56 | 340
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 77 | 16 | 16 | 109
  White | 182 | 42 | 42 | 266
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 32 | 4 | 4 | 40
  United States | 218 | 53 | 52 | 323
  Australia | 15 | 2 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 5 in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS-10 scale is a clinician-administered questionnaire comprised of 10 items used to measure the severity of MDD symptoms. Scores range from 0 (no apparent symptoms) to 60 (most severe symptoms). Individual questionnaire items include: Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, and Suicidal Thoughts.
Time Frame: Baseline and 5 weeks for each stage
Population: Stage 1 and Stage 2 Full Analysis Sets (FAS) consisted of subjects who were randomized and took at least 1 dose of study drug and had at least 1 postbaseline MADRS-10 assessment in the respective stage.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo S1 | ALKS 5461 0.5mg/0.5mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 0.5mg/0.5mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 256 | 58 | 59 | 54 | 55 | 54
units on a scale | -11.1 (0.67) | -8.4 (1.49) | -13.0 (1.50) | -2.2 (1.08) | -4.8 (1.27) | -3.9 (1.13)
Statistical Analysis 1: Comparison: Placebo S1 vs ALKS 5461 2mg/2mg S1 vs Placebo S2 vs ALKS 5461 2mg/2mg S2; Analysis was conducted for each stage separately and overall efficacy was based on combined stage analysis where stage-specific estimates were combined using pre-specified equal weights. Within each stage ALKS 5461 2mg/2mg was compared to placebo (i.e., ALKS 5461 2mg/2mg S1 vs Placebo S1; and ALKS 5461 2mg/2mg S2 vs Placebo S2. The pre-specified order of hypothesis tests was ALKS 5461 2/2 compared to placebo followed by ALKS 5461 0.5mg/0.5mg compared to placebo; Test type: Superiority; p = 0.109, Mixed Models Analysis — Hypothesis tests were two-sided with an alpha of 0.05. Control of type 1 error inflation due to multiplicity was achieved by pre-specifying a fixed sequence for statistical tests; ALKS 5461 was compared to pbo using stage-specific MMRM for MADRS-10 Change from Baseline. Model-derived estimates were combined using equal weights; Least squares mean difference = -1.8, 95% CI 2-sided [-4.1 to 0.4], Standard Error of Mean 1.14 — Estimates below zero favor ALKS 5461
Statistical Analysis 2: Comparison: Placebo S1 vs ALKS 5461 0.5mg/0.5mg S1 vs Placebo S2 vs ALKS 5461 0.5mg/0.5mg S2; Analysis was conducted for each stage separately and overall efficacy was based on combined stage analysis where stage-specific estimates were combined using pre-specified equal weights. Within each stage ALKS 5461 0.5mg/0.5mg was compared to placebo (i.e., ALKS 5461 0.5mg/0.5mg S1 vs Placebo S1; and ALKS 5461 0.5mg/0.5mg S2 vs Placebo S2). The pre-specified order of hypothesis tests was ALKS 5461 2/2 compared to placebo followed by ALKS 5461 0.5/0.5 compared to placebo; Test type: Superiority; p = 0.975, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.0, 95% CI 2-sided [-2.3 to 2.3], Standard Error of Mean 1.17 — Estimates below zero favor ALKS 5461

2. Secondary Outcome: Proportion of Patients Who Exhibited Treatment Response (MADRS-10)
Description: The proportion of subjects demonstrating MADRS-10 treatment response, defined as a >/= 50% reduction in MADRS-10 score from baseline to the end of the efficacy period (Week 5). The MADRS-10 scale is a measure of the severity of MDD symptoms and includes the following 10 items: Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, and Suicidal Thoughts. Scores range from 0 (no apparent symptoms) to 60 (most severe symptoms).
Time Frame: Baseline and 5 weeks for each stage
Population: Stage 1 Full Analysis Set (FAS) consisted of subjects who took at least 1 dose of study drug and had at least 1 postbaseline assessment of MADRS in Stage 1. Stage 2 FAS consisted of Stage 1 placebo non-responders who entered Stage 2 and who received at least 1 dose of study drug and had at least 1 postbaseline assessment of MADRS in Stage 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo S1 | ALKS 5461 0.5mg/0.5mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 0.5mg/0.5mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 256 | 58 | 59 | 54 | 55 | 54
Participants
  Yes | 79 | 9 | 20 | 6 | 9 | 9
  No | 177 | 49 | 39 | 48 | 46 | 45

3. Secondary Outcome: Remission Rate
Description: The proportion of subjects achieving remission, defined as a MADRS-10 score of </= 10 at the end of the efficacy period.
Time Frame: Baseline and 5 weeks for each stage
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo S1 | ALKS 5461 0.5mg/0.5mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 0.5mg/0.5mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 256 | 58 | 59 | 54 | 55 | 54
Participants
  Yes | 47 | 6 | 13 | 4 | 7 | 7
  No | 209 | 52 | 46 | 50 | 48 | 47

4. Secondary Outcome: Number of Subjects With Adverse Events (AEs)
Time Frame: 5 weeks for Stage 1 and 6 weeks for Stage 2
Population: Safety population consists of all randomized subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo S1 | ALKS 5461 0.5mg/0.5mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 0.5mg/0.5mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 265 | 59 | 60 | 56 | 56 | 56
Participants | 142 | 34 | 41 | 29 | 27 | 29

ADVERSE EVENTS:
Time Frame: 5 weeks for Stage 1 and 6 weeks for Stage 2
Description: Safety population consists of all randomized subjects who received at least 1 dose of study drug.
Arm/Group | Placebo S1 | ALKS 5461 0.5mg/0.5mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 0.5mg/0.5mg S2 | ALKS 5461 2mg/2mg S2
All-Cause Mortality (participants affected / at risk) | 0/265 | 0/59 | 0/60 | 0/56 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 1/265 | 0/59 | 0/60 | 0/56 | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 81/265 | 32/59 | 36/60 | 11/56 | 13/56 | 22/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo S1 (N=265) | ALKS 5461 0.5mg/0.5mg S1 (N=59) | ALKS 5461 2mg/2mg S1 (N=60) | Placebo S2 (N=56) | ALKS 5461 0.5mg/0.5mg S2 (N=56) | ALKS 5461 2mg/2mg S2 (N=56)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo S1 (N=265) | ALKS 5461 0.5mg/0.5mg S1 (N=59) | ALKS 5461 2mg/2mg S1 (N=60) | Placebo S2 (N=56) | ALKS 5461 0.5mg/0.5mg S2 (N=56) | ALKS 5461 2mg/2mg S2 (N=56)
Nausea (Gastrointestinal disorders) | 17 (17) | 14 (15) | 17 (24) | 1 (1) | 5 (6) | 8 (8)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4) | 10 (10) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4) | 6 (6) | 0 (0) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 2 (2) | 5 (6) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 5 (5) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (7) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 9 (10) | 4 (4) | 8 (9) | 1 (2) | 4 (4) | 2 (2)
Somnolence (Nervous system disorders) | 7 (7) | 5 (5) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 22 (23) | 7 (10) | 5 (5) | 1 (1) | 1 (1) | 2 (2)
Sedation (Nervous system disorders) | 3 (3) | 2 (2) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 7 (7) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.